CLINICAL TRIAL: NCT04875013
Title: Efficacy of Vestibular Rehabilitation Using Computerized Dynamic Posturography With Virtual Reality for Stable Unilateral Vestibular Weakness
Brief Title: Interactive Rehabilitation for Adults With Unilateral Vestibular Weakness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eytan A. David (Other)
Responsible Party: Sponsor-Investigator, Eytan A. David, MD, FRCSC, Clinical Instructor, Dept. of Surgery, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H20-04045
Record Dates: First submitted 2021-04-27; First posted 2021-05-06 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-11

CONDITIONS: Dizziness; Equilibrium; Disorder, Labyrinth; Inner Ear Injury
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Intervention Model Description: Longitudinal cohort; single group assignment; interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Vestibular rehabilitation with dynamic posturography (Experimental): 12 sessions, twice per week, of rehabilitation exercises last about 20 minutes, using CDP and interactive visual feedback
  Interventions: Device: Vestibular rehabilitation with dynamic posturography

INTERVENTIONS:
Device: Vestibular rehabilitation with dynamic posturography — Rehabilitation exercises guided by an interactive display and measured by a footplate sensor

SUMMARY:
People that have difficulty with balance, such as those with damage to their inner ear, have a higher risk of falling, which may lead to anxiety and reduced quality of life. Some individuals that have lost part of their sense of balance can learn to compensate using information from their vision, their sense of where their limbs are in space, and from other balance organs that are still intact. Our study aims to determine if virtual reality used together with information from footplate sensors can be used to train people with balance problems to compensate for their inner ear deficits.

ELIGIBILITY:
Inclusion Criteria:

* Adult Age 18-80
* Unilateral vestibular weakness confirmed one or more of:

  * Videonystagmography
  * VEMP
* Or unilateral vestibular weakness idiopathic, not yet diagnosed (NYD)
* Persistent imbalance following diagnosis of resolved benign paroxysmal positional vertigo (BPPV)
* Symptomatic
* Long-standing/persistent symptoms greater than one year

Exclusion Criteria:

* Orthopedic deficit (eg. lower body joint dysfunction or lower joint replacement)
* Neurological deficit or proprioception deficit
* Diabetes
* Poor vision or blindness
* Fluctuating vestibular symptoms, or condition known to fluctuate eg. Menière's disease, perilymphatic fistula (PLF) or superior canal deshicsence (SDCS)
* Active benign paroxysmal positional vertigo (BPPV)
* Undergoing treatment which may affect balance or ability to stand
* Cognitive impairment that prevents understanding and responding to instructions required to complete the study
* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eytan David, MD, Principal Investigator — University of British Columbia
Locations (1):
- Dr. EA David MD FRCSC, North Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.

REFERENCES:
- [Derived] David EA, Shahnaz N. Posturographic sensory ratios provide evidence for neuroplasticity after computerized vestibular rehabilitation therapy in a single group interventional trial. J Neuroeng Rehabil. 2025 Apr 11;22(1):81. doi: 10.1186/s12984-025-01608-w. PMID 40217271
- [Derived] David EA, Shahnaz N, Wiseman I, David Y, Cochrane CL. Computerized Dynamic Posturography-Guided Vestibular Rehabilitation Improves Vestibular Sensory Ratios. Ear Nose Throat J. 2025 Mar 12:1455613251321978. doi: 10.1177/01455613251321978. Online ahead of print. PMID 40072844
- [Derived] David EA, Shahnaz N. Dynamic posturography after computerized vestibular retraining for stable unilateral vestibular deficits. Acta Otolaryngol. 2023 May;143(5):396-401. doi: 10.1080/00016489.2023.2208615. Epub 2023 May 12. PMID 37173291
- [Derived] David EA, Shahnaz N. Patient-Reported Disability After Computerized Posturographic Vestibular Retraining for Stable Unilateral Vestibular Deficit. JAMA Otolaryngol Head Neck Surg. 2022 May 1;148(5):426-433. doi: 10.1001/jamaoto.2022.0167. PMID 35357406

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vestibular Rehabilitation With Dynamic Posturography
Started | 13
Post-treatment Assessment | 13
Completed | 9
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Vestibular Rehabilitation With Dynamic Posturography
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 51 [18 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Sensory Organization Test (SOT) Composite Score (Score After Retraining Minus Score at Baseline)
Description: Change in composite score of Sensory Organization Test (SOT) (Scores from 0-100; higher scores indicate better function); Lower scores indicate larger amount of sway
  Calculated as a composite of the 6 individual conditions of the SOT:
  1. Eyes open on firm surface
  2. Eyes closed on firm surface
  3. Eyes open with sway referenced visual
  4. Eyes open on sway referenced support surface
  5. Eyes close on sway referenced support surfrace
  6. Eyes open on sway referenced support surface and visual
Time Frame: Through study completion, 12 rehabilitation sessions, an average of 7 weeks
Measure: Median (95% Confidence Interval); unit: SOT composite score
Arm/Group | Vestibular Rehabilitation With Dynamic Posturography
Number analyzed (Participants) | 13
SOT composite score | 8.8 [0.6 to 19.1]

2. Primary Outcome: Change in Dizziness Handicap Inventory Score (Score After Retraining Minus Score at Baseline)
Description: Change in Dizziness Handicap Inventory (DHI); scale from 0-100; higher scores indicate greater disability; 16-34 Points (mild handicap), 36-52 Points (moderate handicap), 54+ Points (severe handicap)
Time Frame: Through study completion, 12 rehabilitation sessions, an average of 7 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Vestibular Rehabilitation With Dynamic Posturography
Number analyzed (Participants) | 13
score on a scale | -16 [-20 to 2]

3. Primary Outcome: Change in Activities-specific Balance Confidence Scale Score (Score After Retraining Minus Score at Baseline)
Description: Change in Activities-specific Balance Confidence (ABC) score; (Scores from 0-100; higher scores indicate greater confidence in performing activities of daily living)
Time Frame: Through study completion, 12 rehabilitation sessions, an average of 7 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Vestibular Rehabilitation With Dynamic Posturography
Number analyzed (Participants) | 13
score on a scale | 11.87 [0 to 17.30]

4. Primary Outcome: Change in Fall Efficacy Scale-International (FES-I) (Score After Retraining Minus Score at Baseline)
Description: Change in Fall Efficacy Scale-International (FES-I); possible scores 16-64, higher score indicates greater perceived fall risk
Time Frame: Through study completion, 12 rehabilitation sessions, an average of 7 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Vestibular Rehabilitation With Dynamic Posturography
Number analyzed (Participants) | 13
score on a scale | -9 [-14 to 1]

5. Primary Outcome: Change in Limits of Stability Area (Area After Retraining Minus Area at Baseline)
Description: Change in endpoint excursion and maximum excursion functional stability region area, calculated from Limits of Stability (LOS) score Higher score indicates an ability to volitionally lean to larger angles. 100% of theoretical maximum in all directions would give an area of 28284.
  LOS excursion scores were calculated by the instrument software, from which we calculated the area of the endpoint excursion functional stability region (the sum of areas between adjacent Endpoint Excursion limits) and the area of the maximum excursion functional stability region (the sum of areas between adjacent Maximum Excursion limits) using published methods (Alvarez-Otero R, Perez-Fernandez N. The limits of stability in patients with unilateral vestibulopathy. Acta Oto-laryngol. 2017;137(10):1-6. doi:10.1080/00016489.2017.1339326)
Time Frame: Through study completion, 12 rehabilitation sessions, an average of 7 weeks
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Vestibular Rehabilitation With Dynamic Posturography
Number analyzed (Participants) | 13
units on a scale
  Endpoint excursion functional stability region | 6226 [24 to 14547]
  Maximum excursion functional stability region | 9802 [2248 to 21168]

6. Secondary Outcome: Change in Sensory Organization Test Scores for Conditions 1 to 6 (Scores After Retraining Minus Scores at Baseline)
Description: Change in mean Sensory Organization Test Scores for conditions 1 through 6; (Scores from 0-100; higher scores indicate better function)
  The 6 conditions are:
  1. Eyes open on firm surface
  2. Eyes closed on firm surface
  3. Eyes open with sway referenced visual
  4. Eyes open on sway referenced support surface
  5. Eyes close on sway referenced support surfrace
  6. Eyes open on sway referenced support surface and visual
Time Frame: Through study completion, 12 rehabilitation sessions, an average of 7 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Vestibular Rehabilitation With Dynamic Posturography
Number analyzed (Participants) | 13
score on a scale
  SOT condition 1 | 0.6 [-1.5 to 4.3]
  SOT condition 2 | -1.8 [-4.2 to 2.0]
  SOT condition 3 | -1.6 [-3.2 to 2.6]
  SOT condition 4 | 13.9 [3.0 to 27.8]
  SOT condition 5 | 11.1 [1.6 to 23.4]
  SOT condition 6 | 13.1 [2.9 to 34.4]

7. Secondary Outcome: Change in Sensory Organization Test Vestibular Contribution (Ratio After Retraining Minus Ratio at Baseline)
Description: Change in mean value of Sensory Organization Test condition 5/mean value of SOT conditions 1; measured as a ratio, higher scores indicate a greater vestibular contribution to balance deficit
Time Frame: Through study completion, 12 rehabilitation sessions, an average of 7 weeks
Measure: Median (95% Confidence Interval); unit: ratio of scores on a scale
Arm/Group | Vestibular Rehabilitation With Dynamic Posturography
Number analyzed (Participants) | 13
ratio of scores on a scale | 0.10 [-0.06 to 0.25]

8. Secondary Outcome: Change in Limits of Stability Directional Control Component (Score After Retraining Minus Score at Baseline)
Description: Limits of Stability test mean value of directional control of limits of stability; (Scores from 0-100; higher scores indicate better function)
Time Frame: Through study completion, 12 rehabilitation sessions, an average of 7 weeks
Measure: Median (95% Confidence Interval); unit: Directional control %
Arm/Group | Vestibular Rehabilitation With Dynamic Posturography
Number analyzed (Participants) | 13
Directional control % | 41.1 [5.9 to 79]

9. Secondary Outcome: Change in Endpoint and Maximum Excursion Values From Limits of Stability Test (Score After Retraining Minus Score at Baseline)
Description: Limits of Stability test mean endpoint excursion value and maximum excursion point; (Scores from 0-100; higher scores indicate better function)
Time Frame: Through study completion, 12 rehabilitation sessions, an average of 7 weeks
Measure: Median (95% Confidence Interval); unit: excursion as % of limit of stability
Arm/Group | Vestibular Rehabilitation With Dynamic Posturography
Number analyzed (Participants) | 13
excursion as % of limit of stability
  Endpoint excursion | 36 [2 to 51]
  Maximum excursion | 47 [5.9 to 79]

10. Other Pre Specified Outcome: Adherence to Rehabilitation Protocol
Description: Percentage of subjects that complete 12 sessions
Time Frame: Through study completion, maximum of 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vestibular Rehabilitation With Dynamic Posturography
Number analyzed (Participants) | 13
Participants | 13

11. Other Pre Specified Outcome: Missed Sessions
Description: Mean number of missed and rescheduled rehabilitation sessions
Time Frame: Through study completion, maximum of 12 weeks
Measure: Mean (Full Range); unit: number is missed sessions / participant
Arm/Group | Vestibular Rehabilitation With Dynamic Posturography
Number analyzed (Participants) | 13
number is missed sessions / participant | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Duration of the treatment period until the post-treatment follow up (approximately 7 weeks)
Arm/Group | Vestibular Rehabilitation With Dynamic Posturography
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT04875013/Prot_SAP_000.pdf